## **Informed Consent Form**

## Official Study Title: Electronic Device Implantation Through Remote Guidance Unique Protocol ID: #224 NCT Number: NCT06404021 Document Type: Study Protocol and Statistical Analysis Plan Document Date: 17 June 2021 Version: 1.0

## **INFORMED CONSENT FORM**

Informed consent form for participation in the research project " Electronic Device Implantation Through Remote Guidance"

- PURPOSE OF THE STUDY: Implantable cardioverter defibrillators (ICDs) and cardiac resynchronization therapy defibrillators (CRT-Ds) are essential tools for managing patients at risk of life-threatening arrhythmias and heart failure. This study aims to evaluate the feasibility and safety of performing these implantations under remote guidance by a biomedical engineer (Field Clinical Specialist FCS) through a dedicated telemedicine system. The main objectives are: to compare the procedural duration and outcomes between remote and standard FCS support; to assess any differences in fluoroscopy time, device functionality, and adverse events; and to confirm the reliability of device parameters at follow-up.
- PROCEDURES: This is a prospective, randomized pilot study conducted at the "Magna Graecia" University and at University Hospital "Annunziata" of Cosenza. Patients undergoing ICD or CRT-D implantation will be randomly assigned to a procedure with an on-site or remote FCS. The procedure will follow standard protocols, with real-time audiovisual communication guiding the steps of device implantation and programming. There are no additional risks to patients compared to standard procedures.
- CONFIDENTIALITY: Data will be processed in accordance with Article 13 of EU Regulation 2016/679 (GDPR) and the relevant Italian legislation. The Data Controller is the Cardiology Department of the University of Calabria. All data will be collected anonymously and used exclusively for scientific research purposes. Participant anonymity will be ensured by restricting data access to authorized research staff only.
- VOLUNTARY PARTICIPATION AND RIGHT TO WITHDRAW: Participation in this study is entirely voluntary. You have the right to refuse participation or withdraw at any time without giving any reason. There will be no consequences for your medical care.
- DISSEMINATION OF RESULTS: The results of this study will be published in scientific journals and/or presented at national and international conferences. At the end of the study, participants may request access to study results from the investigators or attend a dedicated dissemination session.
- ETHICS COMMITTEE APPROVAL: This study has been approved by the Ethics Committee of the Cardiology Department of the University of Calabria.

| By signing this form, I do | eclare: | |
|---|---|---|
| - That I have read this do | ocument carefully; | |
| - That I have been inforr | ned about the purpo | se and objectives of the study; |
| - That I have had the opp | portunity to ask que | stions and received clear answers; |
| - That I have received su<br>collected during the stud | · · | on the confidentiality of the information |
| - That I am aware I can v | withdraw at any time | 2; |
| - That I freely give my co | onsent to participate | in this study. |
| Date: | Partic | cipant's signature: |
| I, the undersigned, decla | nre: | |
| - That I have received co<br>sheet; | omplete and clear inf | formation and understood the information |
| - That I have had the opp | portunity to ask que | stions and received satisfactory answers; |
| I acknowledge that: | | |
| - Participation in the stu | dy is entirely volunt | ary; |
| - I am free to withdraw a | at any time without j | ustification; |
| - The study has been app | proved by the Ethics | Committee; |
| - Data will be handled in | compliance with EU | J Regulation No. 679/2016. |
| Therefore, I DECLARE: | | |
| ☐ I wish to participate | e in the study | $\square$ I do not wish to participate in the study |

| Full name in block letters | Participant's signature | Date |
|---|---|---|
| Impartial witness (if applicable) | Participant's signature | Date |
| (only if the patient is unable to write | te) | |
| <b>DECLARATION OF THE INVESTI</b> I declare that I have provided the p nature, objectives, procedures, and | atient with full and detailed ex | |
| I also declare that I have given the poops of this Informed Consent Form | | nd a signed and dated |
| Investigator's full name (block lette | ers) Signature | Date |